CLINICAL TRIAL: NCT00015808
Title: Phase I Clinical Trial to Establish the Maximum Tolerated Dose of Idebenone in Children, Adolescents, and Adults With Friedreich's Ataxia
Brief Title: Safety Study of Idebenone to Treat Friedreich's Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010167; 01-N-0167
Record Dates: First submitted 2001-05-06; First posted 2001-05-07 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-04

CONDITIONS: Friedreich Ataxia
Keywords: Neurodegeneration; Anti-Oxidant; Neuropathy; Hereditary; Spinocerebellar; Friedreich's Ataxia; Friedreich Ataxia; FRDA
MeSH Terms: conditions — Friedreich Ataxia; Nerve Degeneration | interventions — idebenone

INTERVENTIONS:
Drug: Idebenone

SUMMARY:
This study will determine the highest dose of idebonone that can safely be given to patients with Friedrich's ataxia, an inherited degenerative disease that causes loss of muscle coordination, speech problems, weakness and sensory loss. Enlargement of the left ventricle (the large pumping chamber of the heart) is also common in this disease. In studies in France and Canada, patients with Friedrich's ataxia who were given idebonone, an antioxidant similar to the dietary supplement coenzyme Q, had a decrease in the size of their left ventricle.

Patients 5 years and older with Friedrich's ataxia may be eligible for this study. Pregnant and lactating women may not participate. Candidates will be screened with a medical history and physical examination and a review of genetic studies. Patients who have not had genetic studies will be offered genetic counseling and testing to confirm or rule out Friedrich's ataxia.

Participants will be admitted to the NIH Clinical Center for 3 days. They will have blood and urine tests and a heart evaluation, including an echocardiogram-a procedure that uses sound waves to produce images of the heart, and an electrocardiogram-a study of the electrical activity of the heart. When these tests have been completed, patients will take an idebonone capsule. They will be monitored for side effects for 72 hours. Blood samples will be collected through an intravenous catheter (flexible plastic tube placed in a vein) 0.5, 1, 2, 3, 4, 6, 12, 24, 48 and 72 hours after the drug is taken to determine how long it takes for the drug to be eliminated from the body.

Patients will return for a follow-up visit within 1 to 8 weeks. Those who experienced no serious side effects may receive another, higher dose of the drug, with at least 6 days between doses.

DETAILED DESCRIPTION:
Friedreich's ataxia (FRDA) is a progressive, autosomal recessive, multisystem degenerative disease for which there is currently no effective treatment. Recent studies suggest that lipid-soluble antioxidants may prevent the progression of neurodegeneration and lead to some reversal of cardiomyopathy.

This will be a phase Ia, unblinded, dose-escalation trial examining the toxicity and tolerability of the antioxidant idebenone in patients with FRDA. Our primary objective is to determine the maximum tolerated single dose of idebenone in patients with FRDA. Our secondary objective is to document the pharmacokinetics of single-dose idebenone in this population. We aim to enroll 48 patients divided evenly among three age cohorts: children (ages 5-11), adolescents (ages 12-17), and adults (age greater than or equal to 18). Each age cohort will be studied independently. Three patients from each cohort will receive one day of oral idebenone followed by inpatient monitoring for 72 hours. If dose-limiting toxicity (DLT) is not observed during the 72-hour study period, three new patients will receive the next highest dose. If one of three patients experiences DLT, three new patients will receive the same dose. Within each cohort, the dose will be escalated until the maximum tolerated dose (MTD) is established. The MTD will be defined as one dose below that which resulted in DLT in any two patients within a cohort.

Subsequent to the completion of this phase Ia trial, we plan to further refine the MTD for each age group in a phase Ib trial in which we will examine multiple-dose regimens over a longer study period. We hope to follow these phase I studies with a double-blinded, placebo-controlled phase II trial to further evaluate safety and to estimate the efficacy of idebenone using cardiac parameters as our primary endpoints. In addition, we are currently in the process of validating a clinical evaluation scale for FRDA that we hope to employ in measuring neurological parameters as a secondary endpoint in the phase II trial.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of FRDA with confirmed FRDA mutations.

Age greater than or equal to five years old.

No exposure to idebenone or coenzyme Q10 for a period of at least one week prior to onset of the medication phase of the study.

Written, informed consent (and assent, if applicable).

EXCLUSION CRITERIA:

History of a hypersensitivity reaction to idebenone or coenzyme

Q10.

Pregnant or lactating women. All women of child-bearing potential must have negative serum pregnancy prior to the medication phase of the study.

Age less than five years old.

Platelet count, lymphocyte count or hemoglobin below the lower limit of normal.

Alkaline phosphatase, SGOT, SGPT greater than 1.5 times the upper limit of normal. Bilirubin greater than 1.2 g/dl.

Creatinine greater than 1.5 times the upper limit of normal.

Clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2001-05; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Babcock M, de Silva D, Oaks R, Davis-Kaplan S, Jiralerspong S, Montermini L, Pandolfo M, Kaplan J. Regulation of mitochondrial iron accumulation by Yfh1p, a putative homolog of frataxin. Science. 1997 Jun 13;276(5319):1709-12. doi: 10.1126/science.276.5319.1709. PMID 9180083
- [Background] Beal MF. Energetics in the pathogenesis of neurodegenerative diseases. Trends Neurosci. 2000 Jul;23(7):298-304. doi: 10.1016/s0166-2236(00)01584-8. PMID 10856939
- [Background] Campuzano V, Montermini L, Molto MD, Pianese L, Cossee M, Cavalcanti F, Monros E, Rodius F, Duclos F, Monticelli A, Zara F, Canizares J, Koutnikova H, Bidichandani SI, Gellera C, Brice A, Trouillas P, De Michele G, Filla A, De Frutos R, Palau F, Patel PI, Di Donato S, Mandel JL, Cocozza S, Koenig M, Pandolfo M. Friedreich's ataxia: autosomal recessive disease caused by an intronic GAA triplet repeat expansion. Science. 1996 Mar 8;271(5254):1423-7. doi: 10.1126/science.271.5254.1423. PMID 8596916
- [Derived] Di Prospero NA, Sumner CJ, Penzak SR, Ravina B, Fischbeck KH, Taylor JP. Safety, tolerability, and pharmacokinetics of high-dose idebenone in patients with Friedreich ataxia. Arch Neurol. 2007 Jun;64(6):803-8. doi: 10.1001/archneur.64.6.803. PMID 17562928